CLINICAL TRIAL: NCT01952275
Title: Assessment of the Enrichment of Rare Coding Genetic Variants in Patients Affected by Neutrophil-Mediated Inflammatory Dermatoses
Brief Title: Observational Study of the Genetic Architecture of Neutrophil-Mediated Inflammatory Skin Diseases
Acronym: NEUTROGENE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: USZ-DER-AAN-019
Record Dates: First submitted 2013-09-17; First posted 2013-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Other Specified Inflammatory Disorders of Skin or Subcutaneous Tissue; Pyoderma Gangrenosum; Erosive Pustular Dermatosis of the Scalp; Sweet's Syndrome; Behcet's Disease; Bowel-associated Dermatosis-arthritis Syndrome; Pustular Psoriasis; Acute Generalized Exanthematous Pustulosis; Keratoderma Blenorrhagicum; Sneddon-Wilkinson Disease; IgA Pemphigus; Amicrobial Pustulosis of the Folds; Infantile Acropustulosis; Transient Neonatal Pustulosis; Neutrophilic Eccrine Hidradenitis; Rheumatoid Neutrophilic Dermatitis; Neutrophilic Urticaria; Still's Disease; Erythema Marginatum; Unclassified Periodic Fever Syndromes / Autoinflammatory Syndromes; Dermatitis Herpetiformis; Linear IgA Bullous Dermatosis; Bullous Systemic Lupus Erythematosus; Inflammatory Epidermolysis Bullosa Aquisita; Neutrophilic Dermatosis of the Dorsal Hands (Pustular Vasculitis); Small Vessel Vasculitis Including Urticarial Vasculitis; Erythema Elevatum Diutinum; Medium Vessel Vasculitis
MeSH Terms: conditions — Pyoderma Gangrenosum; Sweet Syndrome; Behcet Syndrome; Acute Generalized Exanthematous Pustulosis; Keratosis; Skin Diseases, Vesiculobullous; Hidradenitis; Arthritis, Juvenile; Dermatitis Herpetiformis; Linear IgA Bullous Dermatosis; Erythema elevatum diutinum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva or Blood Serum Histology FFPE
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Collection of biological samples

SUMMARY:
This study investigates the genetic architecture of Neutrophil-Mediated Inflammatory Skin Diseases. After collecting informed consent, all patients' clinical phenotype is graded at inclusion with a detailed case report form and a discovery cohort formed based on the certainty of diagnosis. The DNA of patients in the discovery cohort is analyzed by whole exome sequencing which identifies all protein-coding genetic variants. Subsequently, statistical burden tests are going to identify enrichment of rare coding genetic variants in patients affected by Neutrophil-Mediated Inflammatory Skin Diseases.

The ultimate goal is to reveal the responsible gene(s) that may then be targets for clinical intervention.

DETAILED DESCRIPTION:
Timeframe:

* Collection of DNA for discovery cohort until 05/2016
* Data analysis until 12/2014 for pyoderma gangrenosum, until 12/2016 for other NMID
* Report and data presentation early 2015 for PG, 2017 for other NMID

ELIGIBILITY:
Inclusion criteria:

* History of NMID or active disease.
* Informed consent.

Exclusion criteria:

- No consent to either part of the study.

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a history of Neutrophil-Mediated Inflammatory Dermatoses (NMID) of any subtype
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Enrichment of rare coding genetic variants | baseline
  Whole exome sequencing is going to detect rare coding genetic variants in cases of Neutrophil-Mediated Inflammatory Skin Diseases. Statistical burden tests are applied to test for excess of rare variants in cases versus available controls of matching ancestry.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Navarini, MD, Principal Investigator — University Hospital Zurich, Dept. of Dermatology
Locations (1):
- University Hospital Zurich, Dept. of Dermatology, Zurich, Canton of Zurich, Switzerland